CLINICAL TRIAL: NCT05404165
Title: Relevance of the Self-assessment of Skills for Self-administration of Adrenaline by Auto-injectors in Patients at Risk of Severe Anaphylactic Reaction
Brief Title: Relevance of the Self-assessment of Skills for Self-administration of Adrenaline by Auto-injectors in Patients at Risk of Severe Anaphylactic Reaction (PacAdré)
Acronym: PacAdré
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC22.0156
Record Dates: First submitted 2022-05-30; First posted 2022-06-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Severe Anaphylactic Reaction, Self-administration, Adrenaline, Self-assessment
Keywords: Adrenaline; Self-administration; Self-assessment; Severe anaphylactic reaction
MeSH Terms: conditions — Anaphylaxis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To investigate the correlation between self-assessment by patients and an assessment by a health professional of the skills needed for self administration of adrenaline by auto-injectors. These skills include the identification of situations requiring the administration of adrenaline and the technical abilities to achieve it.

Hypothesis:

A self-assessment correlated with an external assessment would make it easier to adjust the frequency of therapeutic education sessions based on the patient's self-assessment alone.

DETAILED DESCRIPTION:
Intramuscular Adrenaline is the standard treatment for severe to moderate anaphylaxis. Self-administration of Adrenaline by the patient using an auto-injector pen in case of anaphylaxis is a major axis of management of patients with severe food allergy, hymenoptera venom allergy or systemic mastocytosis. This self-administration skill requires prior therapeutic education of the patient. This education must be repeated over time and must include two components: the identification of anaphylactic situations requiring the self-administration of Adrenalin and the technical skills and abilities to carry out this self-injection.

Numerous studies have investigated the technical skills for using Adrenaline auto-injector pens according to the device prescribed, the importance of therapeutic education, the optimal frequency of therapeutic education sessions for self-administration and the main barriers to the use of Adrenaline.

To our knowledge, no study has investigated the correlation between patients' self-assessment of the skills required for self-administration of Adrenaline by self-injecting pen and an external assessment of these same skills by a health professional.

A self-assessment correlated with an external assessment would make it easier to adjust the frequency of therapeutic education sessions based on patient self-assessment alone.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Follow-up at the CHU Grenoble Alpes or at the CH Métropole Savoie with at least one consultation every 2 years
* With a pathology at risk of severe anaphylaxis:

  * Severe food allergy and/or,
  * Allergy to wasp venom and/or
  * Systemic mastocytosis
* With a current adrenaline prescription that is more than a year old

Exclusion Criteria:

* Patient with a pathology at risk of severe anaphylaxis not identified in the inclusion criteria (isolated drug allergy, idiopathic anaphylaxis, etc.)
* Patient with cognitive or memory disorders
* Patient not speaking French or with a limited understanding of the language
* Patient not affiliated to a social security scheme
* Refusal of the patient to participate in the research or inability of the patient to give his consent
* Patient under guardianship or subject deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are being monitored for severe allergy or systemic mastocytosis and who need to have adrenaline treatment with them in case of anaphylaxis.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2022-05-23 (Estimated); Primary Completion 2022-08-15 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between a patient self-assessment and a health care professional's assessment of the skills needed to self-administer epinephrine by self-injecting pen | One day
  A two-part, 20-point self-assessment scale:
  * A visual analog scale addressing skills in identifying situations requiring administration of self-injectable epinephrine, scored out of 10 points
  * A visual analogue scale for technical skills in administering epinephrine by self-injecting pen, scored out of 10 points
  A two-part health professional assessment scale scored out of 20 points:
  * A single response questionnaire asked to the patient including 5 standardized clinical situations, validated by an expert committee, requiring or not the administration of Adrenalin, scored out of 10 points
  * An evaluation of the technical skills of injecting adrenaline with a self-injecting pen with a demonstration pen, in 6 steps, scored out of 10 points

SECONDARY OUTCOMES:
Correlation between patient self-assessment and healthcare professional assessment of ability to identify situations requiring administration of self-injectable epinephrine | One day
  A 10-point self-assessment scale in the form of a visual analogue scale on the ability to identify situations requiring the administration of self-injectable epinephrine and a hetero-assessment with a 10-point single-answer questionnaire including 5 standardized clinical situations, validated by an expert committee, requiring or not the administration of adrenaline
Correlation between a patient's self-assessment and a healthcare professional's assessment of technical skills in performing epinephrine administration by self-injecting pen | One day
  A 10-point self-assessment scale in the form of a visual analog scale of technical skills in performing epinephrine administration by self-injecting pen and a 10-point hetero-assessment of epinephrine injection skills by self-injecting pen with a 6-step demonstration pen.

CONTACTS AND LOCATIONS:
Overall Officials: Alexis BOCQUET, Md, Principal Investigator — CHU Grenoble Alpes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bilo MB, Cichocka-Jarosz E, Pumphrey R, Oude-Elberink JN, Lange J, Jakob T, Bonadonna P, Fernandez J, Kosnik M, Helbling A, Mosbech H, Gawlik R, Niedoszytko M, Patella V, Pravettoni V, Rodrigues-Alves R, Sturm GJ, Rueff F. Self-medication of anaphylactic reactions due to Hymenoptera stings-an EAACI Task Force Consensus Statement. Allergy. 2016 Jul;71(7):931-43. doi: 10.1111/all.12908. Epub 2016 Apr 29. PMID 27060567
- [Background] Muraro A, Werfel T, Hoffmann-Sommergruber K, Roberts G, Beyer K, Bindslev-Jensen C, Cardona V, Dubois A, duToit G, Eigenmann P, Fernandez Rivas M, Halken S, Hickstein L, Host A, Knol E, Lack G, Marchisotto MJ, Niggemann B, Nwaru BI, Papadopoulos NG, Poulsen LK, Santos AF, Skypala I, Schoepfer A, Van Ree R, Venter C, Worm M, Vlieg-Boerstra B, Panesar S, de Silva D, Soares-Weiser K, Sheikh A, Ballmer-Weber BK, Nilsson C, de Jong NW, Akdis CA; EAACI Food Allergy and Anaphylaxis Guidelines Group. EAACI food allergy and anaphylaxis guidelines: diagnosis and management of food allergy. Allergy. 2014 Aug;69(8):1008-25. doi: 10.1111/all.12429. Epub 2014 Jun 9. PMID 24909706
- [Background] Broesby-Olsen S, Dybedal I, Gulen T, Kristensen TK, Moller MB, Ackermann L, Saaf M, Karlsson MA, Agertoft L, Brixen K, Hermann P, Stylianou E, Mortz CG, Torfing T, Havelund T, Sander B, Bergstrom A, Bendix M, Garvey LH, Bjerrum OW, Valent P, Bindslev-Jensen C, Nilsson G, Vestergaard H, Hagglund H. Multidisciplinary Management of Mastocytosis: Nordic Expert Group Consensus. Acta Derm Venereol. 2016 Jun 15;96(5):602-12. doi: 10.2340/00015555-2325. PMID 26694951
- [Background] Sirin Kose S, Asilsoy S, Tezcan D, Al S, Atay O, Kangalli O, Uzuner N, Karaman O. Is There an Optimal Training Interval to Improve the Correct Use of Adrenaline Auto-Injectors? Int Arch Allergy Immunol. 2020;181(2):136-140. doi: 10.1159/000504365. Epub 2019 Dec 3. PMID 31794965
- [Background] Topal E, Bakirtas A, Yilmaz O, Ertoy IH, Arga M, Demirsoy MS, Turktas I. A real-life study on acquired skills from using an adrenaline autoinjector. Int Arch Allergy Immunol. 2013;160(3):301-6. doi: 10.1159/000341367. Epub 2012 Oct 18. PMID 23095342
- [Background] Ridolo E, Montagni M, Bonzano L, Savi E, Peveri S, Costantino MT, Crivellaro M, Manzotti G, Lombardi C, Caminati M, Incorvaia C, Senna G. How far from correct is the use of adrenaline auto-injectors? A survey in Italian patients. Intern Emerg Med. 2015 Dec;10(8):937-41. doi: 10.1007/s11739-015-1255-z. Epub 2015 May 20. PMID 25990486
- [Background] Segal N, Garty BZ, Hoffer V, Levy Y. Effect of instruction on the ability to use a self-administered epinephrine injector. Isr Med Assoc J. 2012 Jan;14(1):14-7. PMID 22624436
- [Background] Shemesh E, D'Urso C, Knight C, Rubes M, Picerno KM, Posillico AM, Atal Z, Annunziato RA, Sicherer SH. Food-Allergic Adolescents at Risk for Anaphylaxis: A Randomized Controlled Study of Supervised Injection to Improve Comfort with Epinephrine Self-Injection. J Allergy Clin Immunol Pract. 2017 Mar-Apr;5(2):391-397.e4. doi: 10.1016/j.jaip.2016.12.016. Epub 2017 Jan 20. PMID 28117270
- [Background] Song TT, Worm M, Lieberman P. Anaphylaxis treatment: current barriers to adrenaline auto-injector use. Allergy. 2014 Aug;69(8):983-91. doi: 10.1111/all.12387. Epub 2014 May 16. PMID 24835773
- [Background] Simons FE, Ardusso LR, Bilo MB, El-Gamal YM, Ledford DK, Ring J, Sanchez-Borges M, Senna GE, Sheikh A, Thong BY; World Allergy Organization. World Allergy Organization anaphylaxis guidelines: summary. J Allergy Clin Immunol. 2011 Mar;127(3):587-93.e1-22. doi: 10.1016/j.jaci.2011.01.038. No abstract available. PMID 21377030
- [Background] Yu JE, Lin RY. The Epidemiology of Anaphylaxis. Clin Rev Allergy Immunol. 2018 Jun;54(3):366-374. doi: 10.1007/s12016-015-8503-x. PMID 26357949
- [Background] Pumphrey RS. Lessons for management of anaphylaxis from a study of fatal reactions. Clin Exp Allergy. 2000 Aug;30(8):1144-50. doi: 10.1046/j.1365-2222.2000.00864.x. PMID 10931122
- See also: Prise en charge de l'anaphylaxie en médecine d'urgence. — http://www.sfmu.org/upload/consensus/rfe_anaphylaxie_sfmu2016.pdf